CLINICAL TRIAL: NCT06141655
Title: Pragmatic Randomized Trial to Evaluate the Effectiveness of High-Dose Quadrivalent Influenza Vaccine vs. Standard-Dose Quadrivalent Influenza Vaccine in Adults Aged 65 to 79 Years in Galicia, Spain
Brief Title: HD vs SD Quadrivalent Influenza Vaccine in Adults Aged 65 to 79 Years in Galicia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico Martinón Torres (Other)
Responsible Party: Sponsor-Investigator, Federico Martinón Torres, Principal investigator, Hospital Clinico Universitario de Santiago
Organization: Hospital Clinico Universitario de Santiago (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GALFLU
Record Dates: First submitted 2023-10-26; First posted 2023-11-21 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2023-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QIV-HD vaccine (Experimental): EFLUELDA, Suspension for injection, one dose
  Interventions: Drug: Influenza vaccine
- QIV-SD vaccine (Active Comparator): INFLUVAC TETRA, Suspension for injection, one dose
  Interventions: Drug: Influenza vaccine

INTERVENTIONS:
Drug: Influenza vaccine — Participants will be individually randomized 1:1 to receive either QIV-HD or QIV-SD, one dose, the day of the inclusion in the trial

SUMMARY:
This pragmatic randomized trial is designed to evaluate the relative vaccine effectiveness of QIV-HD vs. QIV-SD in reducing the risk of hospitalization for influenza or pneumonia in adults 65-79 years of age in Galicia during 2023/2024 and 2024/2025 seasons.

DETAILED DESCRIPTION:
The study is a pragmatic, registry-based, open-label, active-controlled, individually randomized trial using the infrastructure of the Regional Vaccination Program of Galicia for patient recruitment, inclusion, randomization, and vaccine administration and the Galician health registries for data collection including baseline information, follow-up data and safety monitoring. Participants will have the opportunity of receiving all the information for the trial prior to the vaccination appointment. Informed consent will be obtained during the vaccination appointment by the study team prior to their vaccine administration. The participation in the study is voluntary, and only individuals who accept signing the informed consent will be recruited. Participants may withdraw from the study at any point.

The study aims to randomize at least 114.011 participants over 2 influenza seasons (2023/2024 and 2024/2025) with approximately 57,000 participants per season (pending any further potential sample size adjustments following interim analysis).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 65-79 years residing in the community (only individuals who are not eligible to receive QIV-HD as part of the standard of care)
* 2. Informed consent form has been signed and dated

Exclusion Criteria:

* There are no specific exclusion criteria for this study

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 134476 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of a hospitalization due to influenza or pneumonia | ≥14 days after vaccination and up to May 31 the following year

SECONDARY OUTCOMES:
Hospitalization for any cardio-respiratory disease [composite endpoint] | ≥14 days after vaccination and up to May 31 the following year
All-cause hospitalization | ≥14 days after vaccination and up to May 31 the following year
All-cause mortality | ≥14 days after vaccination and up to May 31 the following year
Hospitalization for influenza | ≥14 days after vaccination and up to May 31 the following year
Hospitalization for pneumonia | ≥14 days after vaccination and up to May 31 the following year

CONTACTS AND LOCATIONS:
Locations (1):
- General Public Health Directorate of Galician Health Service, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pardo-Seco J, Rodriguez-Tenreiro-Sanchez C, Gine-Vazquez I, Mallah N, Miras-Carballal S, Pineiro-Sotelo M, Cribeiro-Gonzalez M, Conde-Pajaro M, Gonzalez-Perez JM, Rivero-Calle I, Bello X, Razzini JL, Dacosta-Urbieta A, Salas A, Harris RC, Loiacono MM, van Aalst R, Farre JM, Dufournet M, Johansen ND, Modin D, Biering-Sorensen T, Duran-Parrondo C, Martinon-Torres F; GALFLU Trial Team. High-Dose Influenza Vaccine to Reduce Hospitalizations. N Engl J Med. 2025 Dec 11;393(23):2303-2312. doi: 10.1056/NEJMoa2509834. Epub 2025 Aug 30. PMID 40888694